CLINICAL TRIAL: NCT02102542
Title: Efficacy of Intravenous Glyco-P® in Patients Undergoing Procedure That Require Anesthesia Service
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Prasert Sawasdiwipachai, Attending physician, Mahidol University
Other Study IDs: 185/2555(EC3)
Record Dates: First submitted 2014-03-30; First posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-03

CONDITIONS: Hypersalivation; Prevention of Drooling; Bradycardia; Reversal of Muscle Relaxants
Keywords: glycopyrrolate; efficacy; antisialagogue
MeSH Terms: conditions — Sialorrhea; Bradycardia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Antisialagouge: A group of patients enrolled to prove efficacy of Glyco-P for reduction of secretions.
- Bradycardia: A group of patients enrolled to prove efficacy of Glyco-P for modest increase of heart rate.
- For reversal of neuromuscular blocking agents: Group of patients enrolled to prove efficacy of Glyco-P when used in combination with neostigmine to reserve neuromuscular blocking agents.

SUMMARY:
This observational study was designed to prove clinical efficacy of the well known "glycopyrrolate" which is considered an orphan drug in Thailand. Since the medication has never been officially used in Thai people and this particular brand "Glyco-P" which was made in India has never been officially proven of its efficacy in Thai people. The study was aimed to prove if this Glyco-P can modestly increase patient's heart rate, decrease secretion and safely used in combination with neostigmine for reversal of non-depo muscle relaxant drugs.

DETAILED DESCRIPTION:
Background and rationale Glycopyrrolate has been long used since it's first discovery in 19602. The medication is generally available in both oral and injectable form. The uses of glycopyrrolate in anesthesia are mainly for reduction of salivation and secretion3, which plays significant role when airway instrumentation required. The widespread uses of neostigmine for reversal of muscle relaxant effects caused by non-depolarizing muscle relaxant also mandate the co-administration of anti-muscarinic4,5,6. Without availability of glycopyrrolate, atropine was used in Thailand, which results in excessive tachycardia and salivation7,8,9. Glycopyrrolate can also be used when mild bradycardia is encountered but the effects on heart rate is less dominant than atropine10,11.

Glycopyrrolate is considered an orphan drugs in Thailand. There was simply no availability until recently. The local company named "Masu" has decided to market and import the drug from India (Glyco-P®). The formulary has been approved by Thai Food and Drug Administration1. The preparation has also been tested in laboratory by third party well-known pharmacy institute, which proved the existence of an active ingredient. However, the uses of this medication officially have not been made and the appropriate action is to obtain IRB approval at local institution and consent the patients prior to drug administration. The appropriate record of clinical effect should also been made.

Objective

1. Evaluate the clinical efficacy of glycopyrrolate on heart rate, anti-sialagogue effects and when used in conjunction with neostigmine for reversal of neuromuscular blockade.
2. Evaluate the timing, onset and duration of glycopyrrolate injection at different dose.

Materials, participants and study method The study requires

1. 100 patients who scheduled to undergo procedure or operation that require anesthesia service who meet criteria for the uses of glycopyrrolate which includes - requirement of anti-sialogogue, mild bradycardia and in whom receiving neostigmine for reversal of neuromuscular blocking agents.
2. Glyco-P injection
3. Monitorings that capable of HR, BP measurement
4. Suctioning equipment with volumetric measurement
5. Clinician evaluating the effects of medication
6. Timer Participants:- 100 adult male or female patients, over 18 year old who consent to the study.

Exclusion Criteria : Children < 18 yo, pregnant or parturient of breast feeding patients, patients who refused or unable to give consent, patients who has co-existing problems with dry secretion i.e. Sjögren's syndrome, glaucoma, myasthenia gravis, patient whom baseline heart rate is > 100 bpm Study method

1. The patient who meet inclusion criteria will be consent to receive medications.
2. The medications will be administered only 1 of these criteria are met

   * To increase heart rate modestly
   * For reduction of secretion or salivation
   * To co-administration with neostigmine
3. The medications will be given in the following fashion

   * Glyco-P 4 mcg/kg IV, repeatedly if no effects. Halt if HR > 100 bpm
   * Glyco-P 0.2 mg per each mg of neostigmine used
4. The clinical effects i.e. heart rate, blood pressure, amount of secretion removed will be recorded along with timing of onset and offset.
5. Collected data will be analyzed by statistician with appropriate statistical methods.

Data analysis

1. Demographic data or each participants
2. Dose and indication of treatment of studied drugs
3. Timing of clinical effects
4. Changes in heart rate and blood pressure
5. Efficacy of reduction of saliva and secretion

Duration of study 3 months Benefit of the study Confirmation of clinical efficacy of this Indian made glycopyrrolate - Glyco-P® in Thai patients.

Other institutions participation None

ELIGIBILITY:
Inclusion Criteria:

* adult over 18 years of age, undergoing procedure that require anesthesia service.
* meet criteria for prevention of drooling, hypersalivation or bradycardia or require reversal of muscle relaxants.

Exclusion Criteria:

* children < 18 years old,
* pregnant or parturient of breast feeding patients,
* patients who refused or unable to give consent,
* patients who has co-existing problems with dry secretion (i.e. Sjögren's syndrome, glaucoma, myasthenia gravis),
* patient whom baseline heart rate is > 100 bpm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants:- 100 adult male or female patients, over 18 year old who consent to the study.
  Exclusion Criteria : Children < 18 yo, pregnant or parturient of breast feeding patients, patients who refused or unable to give consent, patients who has co-existing problems with dry secretion i.e. Sjögren's syndrome, glaucoma, myasthenia gravis, patient whom baseline heart rate is > 100 bpm
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of Glyco-P as an antisialagogue | 3 months
  Examine efficacy of Glyco-P for reduction of secretion and also for prevention of secretion. The secretions score ranges from 0-5 was evaluated by a person who was blinded to treatment before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology Department Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Salem MG, Richardson JC, Meadows GA, Lamplugh G, Lai KM. Comparison between glycopyrrolate and atropine in a mixture with neostigmine for reversal of neuromuscular blockade. Studies in patients following open heart surgery. Br J Anaesth. 1985 Feb;57(2):184-7. doi: 10.1093/bja/57.2.184. PMID 2857570